CLINICAL TRIAL: NCT02126332
Title: A MULTICENTER, RANDOMIZED, CONTROLLED STUDY OF EPIDURAL ANALGESIA FOR SEVERE ACUTE PANCREATITIS
Brief Title: Epidural Analgesia for Pancreatitis (Epipan Study)
Acronym: EPIPAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0188; 2013-004652-37
Record Dates: First submitted 2014-04-11; First posted 2014-04-30 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2014-05

CONDITIONS: Severe Acute Pancreatitis
Keywords: Severe acute pancreatitis; Epidural analgesia; Acute respiratory failure; Mechanical ventilation; Intensive Care Unit (ICU)
MeSH Terms: conditions — Pancreatitis | interventions — Ropivacaine; Sufentanil; Acetaminophen; Nefopam; Tramadol

ARMS (2):
- Conventional group (Other): 2 groups: a " conventional group " in which available guidelines on analgesia are applied, and an " EA " group in which patients receive thoracic EA for at least 3 days.
  Interventions: Other: acetaminophen, nefopam, tramadol, opidoids
- EA group (Epidural anesthesia ) (Experimental): 2 groups: a " conventional group " in which available guidelines on analgesia are applied, and an " EA " group in which patients receive thoracic EA for at least 3 days.
  Interventions: Other: ropivacaine and sufentanil

INTERVENTIONS:
Other: ropivacaine and sufentanil — Thoracic epidural analgesia will be performed using ropivacaine (2 mg/ml), sufentanil (0.5 microg/ml) administered through a patient-controlled deviced (PCEA : patient-controlled epidural analgesia). PCEA parameters will be fixed as follows : continuous administration of 5 to 15 ml/h and bolus of 3 to 10 ml every 10 minutes. Iterative epidural administration of clonidine (1 mckg/kg) will be allowed to achieve analgesia goals.
  Arms: EA group (Epidural anesthesia )
Other: acetaminophen, nefopam, tramadol, opidoids — Conventional analgesia will include enteral and/or parental administration of usual analgesics, ranging from step 1 to step 3 drugs according to WHO classification (including acetaminophen, nefopam, tramadol, opidoids). The route, dose and frequency of analgesics administrations will be based on participating ICUs protocols.
  Arms: Conventional group

SUMMARY:
Acute pancreatitis (AP) is a common disease whose incidence in the US reaches 35 per 100,000 population annually. Its main causes in adults are gallstone migration into the common bile duct and alcohol abuse. Approximately 80% of patients with AP will develop a mild disease for which the management is mainly conservative. However 20% will develop a severe form, which is known to be associated with the development of local complications, such as pancreatic and peripancreatic necrosis, pseudocysts, and systemic complications, such as adult respiratory distress syndrome or renal failure. In the severe form of AP the mortality rate can reach 17% mainly due to multiple organ failure and pancreatic necrosis. In particular, pancreatic necrosis is associated with a death rate of up to 40%.

Epidural anesthesia (EA) is widely used to induce analgesia in the perioperative period and has also been used to decrease pain in patients with AP. In addition, experimental studies have shown a specific beneficial effect of EA in AP, attributed to an anti-inflammatory effect of local anesthetics administered in the epidural space combined with a sympathetic nerve blockade, which redistributes splanchnic blood flow to non-perfused pancreatic regions.

To date, EA has not been adequately tested in intensive care unit (ICU) patients with severe AP, with regards to clinical outcome. The objective of our study is therefore to test the effect of EA on lung dysfunction during severe AP, as we hypothesize that EA could limit lung failure requiring invasive mechanical ventilation (MV) or the duration of invasive MV

DETAILED DESCRIPTION:
BACKGROUND:

Mild acute pancreatitis has a low mortality rate, but patients with severe acute pancreatitis (AP) are more likely to have complications and a much higher death rate. Severe pancreatic injury occurs in 20% of the patients, and 15% to 25% of these patients will not survive. The amplifying effects of inflammatory and oxidative impairment often lead to SAP-induced complications, which are often regarded as hallmarks of severe AP and herald a noted poor outcome. Since respiratory failure is the main cause of death in patients with severe AP, more work is needed for us to prevent and treat AP-associated lung dysfunction Despite recent substantial improvements in the multidisciplinary management of AP (with special emphasis on fluid therapy, intensive care management, prevention of infectious complications, nutritional support, biliary tract management or necrotizing pancreatitis management), the prognosis of severe AP remains poor in patients who develop acute respiratory failure requiring intubation and invasive respiratory support.

Animal studies suggest that epidural analgesia (EA) may decrease the severity of AP. EA is associated with sympathetic nerve blockade, which redistributes splanchnic blood flow to non-perfused pancreatic regions, and it may improve the pancreatic hypoperfusion induced by AP. EA also decreases the severity of metabolic acidosis and tissue injury, thus preventing the progression from an edematous disease to a necrotizing AP.

To date, EA has not been adequately tested in patients with severe AP as compared to conventional management, and with special emphasis on its putative beneficial ventilatory effects.

DESIGN NARRATIVE:

The purpose of this multicenter, prospective, randomized, controlled, trial is to test the effects of thoracic EA on pulmonary outcome in patients with severe AP.

After inclusion, ICU patients with severe AP will be randomized into 2 groups: a " conventional group " in which available guidelines on analgesia are applied, and an " EA " group in which patients receive thoracic EA for at least 3 days. Beyond the analgesic strategy, recent consensual guidelines on the management of severe AP are applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU for acute pancreatitis

Exclusion Criteria:

* Absolute contra-indication for thoracic epidural catheter placement (Prothrombin time < 60%, Platelet count < 75G/l, curative anticoagulant therapy interrupted for less than 8 hours, local infection, active central nervous system infection, history of back surgery associated with a dural space procedure, suspected or confirmed intracranial hypertension, refractory circulatory shock)
* Refractory circulatory shock despite appropriate resuscitation
* Known allergy to ropivacain, sufentanil or clonidine
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days | at day 30
  (defined as the number of days from day 1 to day 30 on which a patient is able to breathe without invasive assistance. A difference in ventilator-free days can reflect a difference in mortality, ventilator days among survivors, or both.)

SECONDARY OUTCOMES:
Duration of invasive and/or non invasive mechanical ventilation | at day 30
incidence of various complications | at day 30
  (death, organ failure, severe sepsis, septic shock, acute respiratory distress syndrome (ARDS), acute respiratory failure, abdominal compartment syndrome, intra- or extra-abdominal infections, pancreatic necrosis or abscess (infected or not), hemodynamic failure requiring vasopressor therapy, acute renal failure, requirement for renal replacement therapy, infected intra-abdominal abscesses requiring drainage (radiological, endoscopic or surgical).
Biological inflammatory response | at inclusion (day 0), on day 2 and day 7
  (biomarker analyses) : plasma levels of interleukin-6, soluble RAGE (receptor for advanced glycation end-products) and neutrophil gelatinase-associated lipocalin (NGAL), urine levels of tissue inhibitor of metalloproteinase 2 (TIMP-2) and insulin-like growth factor binding protein7 (IGFBP-7) (Nephrocheck, Astute Medical)
Cost analysis of severe AP management | at day 30
Incidence of the intolerance to enteral feeding | from inclusion to day 30
Effectiveness of pain management | from day 0 to day 30
  (pain assessment scores : visual analogic scale, behavioral pain scale)
Duration of EA (Epidural anesthesia) therapy | from day 0 to day 30 after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu JABAUDON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jabaudon M, Genevrier A, Jaber S, Windisch O, Bulyez S, Laterre PF, Escudier E, Sossou A, Guerci P, Bertrand PM, Danin PE, Bonnassieux M, Buhler L, Heidegger CP, Chabanne R, Godet T, Roszyk L, Sapin V, Futier E, Pereira B, Constantin JM; EPIPAN study group. Thoracic epidural analgesia in intensive care unit patients with acute pancreatitis: the EPIPAN multicenter randomized controlled trial. Crit Care. 2023 May 31;27(1):213. doi: 10.1186/s13054-023-04502-w. PMID 37259157
- [Derived] Bulyez S, Pereira B, Caumon E, Imhoff E, Roszyk L, Bernard L, Buhler L, Heidegger C, Jaber S, Lefrant JY, Chabanne R, Bertrand PM, Laterre PF, Guerci P, Danin PE, Escudier E, Sossou A, Morand D, Sapin V, Constantin JM, Jabaudon M; EPIPAN Study Group; AzuRea network. Epidural analgesia in critically ill patients with acute pancreatitis: the multicentre randomised controlled EPIPAN study protocol. BMJ Open. 2017 May 29;7(5):e015280. doi: 10.1136/bmjopen-2016-015280. PMID 28554928